CLINICAL TRIAL: NCT04743557
Title: A Phase 1/2, Multicenter, Open-label, Dose-confirmation Trial to Evaluate the Safety and Preliminary Efficacy of DYN101 in Participants 2 to 17 Years of Age With Centronuclear Myopathy Caused by Mutations in MTM1 or DNM2
Brief Title: Early Phase Human Drug Trial to Investigate DYN101 in Participants 2 to 17 Years With Centronuclear Myopathies
Acronym: DyNaMic
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The first Clinical trial with DYN101 (UNITE-CNM) was early terminated. As a consequence, Dynacure decided to not perform this study.
Sponsor: Dynacure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DYN101-C102; 2020-004608-32 (EudraCT Number)
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Centronuclear Myopathy
Keywords: Muscular Diseases; Myopathies, Structural, Congenital; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases
MeSH Terms: conditions — Myopathies, Structural, Congenital; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Weekly infusions of DYN101 at the starting dose level
  Interventions: Drug: DYN101

INTERVENTIONS:
Drug: DYN101 — DYN101, is a constrained ethyl gapmer ASO directed against human DNM2 pre-mRNA

SUMMARY:
There are no available treatments aside from supportive care for patients with Centronuclear myopathy (CNM). This trial will assess the safety and tolerability as well as pharmacokinetics (PK), pharmacodynamics (PD) and preliminary efficacy of DYN101 in participants 2 to 17 years of age with CNM caused by mutations in DNM2 or MTM1.The trial will consist of a pre-screening consent, a screening period, a run-in period (if applicable), and a Part 1 of 12 weeks with weekly infusion of DYN101 to evaluate safety and tolerability as well as PK, PD and preliminary efficacy. The dose level may need adjustment based on the Part 1 results of the current study and available data from the Unite-CNM study (DYN101-C101, NCT04033159). If a dose adjustment is needed, Part 2 will be conducted in the same participants and the newly selected dose level will be used to assess whether efficacy is seen after an additional 12 weeks of treatment. As this trial is investigational, there is no defined, expected benefit for subjects who participate in this trial except a better knowledge of their disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥2 to <18 years on the date the main ICF is signed.
2. Have a clinically symptomatic CNM, with a documented MTM1 or DNM2 mutation.
3. Have impaired muscle function as evidenced by:

   * MFM20 score between 5% and 80% for subjects ≥2 and <6 years of age, or
   * MFM32 score between 5% and 80% for subjects ≥6 years of age.
4. Have sufficient skeletal muscle (vastus lateralis, gastrocnemius, or biceps brachii as last resort) to perform 2 open muscle biopsies during the trial, as determined by ultrasound imaging at screening.
5. Subject must have platelet count >150,000/µL at screening.
6. Parent(s) or legally-authorized representative must be able to provide written, signed and dated informed consent for their child to participate in the trial. Informed assent can be obtained from the child according to local regulations.
7. Parent(s) or legally-authorized representative must be at or above the age of legal consent in the jurisdiction of the country in which the trial is taking place.
8. Subject, parent(s), and/or legally-authorized representative must have an understanding, ability, and willingness to fully comply with visit frequency, trial procedures, videorecording of assessments where applicable, and restrictions, including contraceptive requirements.

Exclusion Criteria:

1. Subject has evidence of clinically significant liver disease.
2. Subject has evidence of clinically significant renal disease.
3. Presence of significant comorbidities or conditions other than CNM or clinically significant findings during screening of medical history, physical examination, clinical laboratory evaluation, vital signs, or ECG recording for which, in the opinion of the investigator and/or the medical monitor, participation would not be in the best interest of the subject (e.g. compromise the safety or well-being) or that could prevent, limit, or confound the protocol-specified assessments (e.g. taking a muscle biopsy).
4. Subject currently enrolled in any interventional trial or scheduled to participate in such a trial whilst participating in the current trial.
5. Subject has previously received gene therapy for CNM.
6. Subject has severe muscle contractures that would preclude the ability to show improvement in the MFM32 assessment, in the opinion of the investigator.
7. Subject has severe airway malacia which could impact the capacity to wean off ventilatory support.
8. Subject requires oxygen supplementation.
9. For female subjects of childbearing potential: pregnant, breastfeeding, or planning to become pregnant during the trial.
10. Current or relevant history of physical or psychiatric illness, and/or any medical disorder that may require treatment or make the subject unlikely to fully complete the trial, or any condition that presents undue risk from the investigational medicinal product (IMP) or procedures.
11. Intake of any disallowed therapies by the subject within 12 weeks before the planned first IMP administration.
12. Known or suspected intolerance or hypersensitivity to IMP ingredients or closely related compounds.
13. Parent(s) or legally authorized representative are legally incapacitated or have limited legal capacity, or have lack of mental capacity to fully understand the protocol requirements and ensure completion of all required trial procedures.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of drug-related Treatment Emergent Adverse Events (TEAEs) | Baseline until Week 12

SECONDARY OUTCOMES:
Measurement of DYN101 concentration in plasma | Week 1 Day 1: before the start of infusion (baseline), immediately after the end of infusion, and at 1, 3, 7, 23, 71 hours after the end of infusion. Week 13 Day 1: predose and 3 hours after the end of infusion
Maximum plasma drug concentration (Cmax) for DYN101 | Week 1 Day 1: before the start of infusion (baseline), immediately after the end of infusion, and at 1, 3, 7, 23, 71 hours after the end of infusion. Week 13 Day 1: predose and 3 hours after the end of infusion
Area under the Plasma Concentration versus Time Curve (AUC) of DYN101 | Week 1 Day 1: before the start of infusion (baseline), immediately after the end of infusion, and at 1, 3, 7, 23, 71 hours after the end of infusion. Week 13 Day 1: predose and 3 hours after the end of infusion

CONTACTS AND LOCATIONS:
Locations (2):
- I-Motion Institute - Trousseau Hospital, Paris, France
- Universitätsklinikum Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tasfaout H, Buono S, Guo S, Kretz C, Messaddeq N, Booten S, Greenlee S, Monia BP, Cowling BS, Laporte J. Antisense oligonucleotide-mediated Dnm2 knockdown prevents and reverts myotubular myopathy in mice. Nat Commun. 2017 Jun 7;8:15661. doi: 10.1038/ncomms15661. PMID 28589938